CLINICAL TRIAL: NCT03682224
Title: A Prospective, Randomized, Single-Blind, Active Control Trial to Compare Safety and Effectiveness Of Liposomal Bupivacaine (Exparel) to Standard Bupivacaine HCl (Marcaine) for Pain Management in Patients Undergoing Video-Assisted Thoracoscopic Lobectomy
Brief Title: Exparel and Marcaine for Pain Management in Thoracoscopic Lobectomy Patients
Acronym: BEMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRABTREE-18-185
Record Dates: First submitted 2018-07-10; First posted 2018-09-24 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer Stage 1
Keywords: clinical trial; bupivacaine-epinephrine; bupivacaine liposome; pain; Morphine equivalent dose; lobectomy; Laproscopic lobectomy; VATS lobectomy; opioid medications
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either Exparel or Marcaine during surgery. Based on the randomization they will receive one of the two drugs. Participants are assigned one of the two groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: The participant will not be aware of the drug group. A study statistician will generate the randomization with two arms. Statistician will be blinded and will not be aware of the treatment allocation. Researchers and clinicians will be aware of the allocation and drugs will be dispensed by the hospital pharmacy based on the allocation sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Active Comparator)
  Interventions: Drug: Liposomal Bupivacaine
- Marcaine (Active Comparator)
  Interventions: Drug: Bupivacaine-Epinephrine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Liposomal Bupivacaine 1.3% (Exparel), 20 ml vial for injection, administered subcutaneously at port site
  Arms: Exparel
Drug: Bupivacaine-Epinephrine — Bupivacaine-Epinephrine 0.25%, 1:200,000 (Marcaine with epinephrine), administered subcutaneously at port site
  Arms: Marcaine

SUMMARY:
The purpose of this study is to assess pain management after elective thoracoscopic lobectomy. The study will compare two local anesthetics that are given intra-operatively during lobectomy to see which one helps in better pain control and to see which one helps decrease the need for opioid medications. Participants will receive either Marcaine (Bupivacaine-epinephrine 0.25%, 1:200,000) or Exparel (Bupivacaine liposomal (1.3%)) and the drug will be chosen in a random fashion. Participants will be followed during the hospital stay and for one year thereafter. An visual Scale will be administered to measure pain, and opioid drug use will be measured by calculating morphine equivalent dose on each day post surgery until discharge and thereafter on 30 day, 6 month and 12 month follow-up visits. Participants will be monitored for any drug related toxicity and other co-morbid conditions for a period on one year post surgery. Overall cost for the surgery and during in hospital stay post surgery will be collected and compared between the two treatment arms.

DETAILED DESCRIPTION:
The hypothesis of this study is the possibility of liposomal bupivacaine providing more relief with less need of narcotics when compared to standard bupivacaine. To test the hypothesis the investigators will compare pain management following local infiltration of liposomal bupivacaine (Exparel®) versus standard bupivacaine HCl with epinephrine (Marcaine®) after VATS (video-assisted thoracoscopic surgery)-lobectomy. This will be accomplished by evaluating total opioid usage and patient reported pain scores.

Study will be conducted at Southern Illinois University-Medicine Clinics and Memorial Medical Center. This is a prospective, randomized, single-blind, active control trial for patients undergoing elective lobectomy. Participants will be randomly assigned to receive either Liposomal Bupivacaine 1.3% or Bupivacaine-Epinephrine 0.25%, 1:200,000 during surgery. Pain management will be monitored via opioid usage and visual pain assessment throughout the hospital stay and at postoperative day 30, 6 month and 1 year follow up visits. Study population includes patients undergoing elective standard of care lobectomy. Based on the power analysis, 150 participants (75 in each randomized group) are required to be enrolled in the study. Taking into consideration a potential loss of 50 participants due to withdrawal, lost to follow up or other reasons, 200 participants will initially be enrolled and randomized to attain 150 participants at the end of study (1-year follow up).

All patients scheduled for surgical consult with Cardiothoracic Surgery for possible video assisted thoracoscopic lobectomy will be screened for initial eligibility criteria. Informed consent form will be discussed in detail at the clinic by authorized study personnel with all participants who are willing to participate in the study. Participants will be given time to review the informed consent with family if so desired. After the participant voluntarily agrees to participate and signs the informed consent form, the inclusion/exclusion criteria will be reviewed again to ensure continued eligibility. Study data including vitals, physical examination, medications, and medical and surgical history will be recorded or obtained from the electronic health records. Participants will be randomly assigned to one of two study drugs- Liposomal Bupivacaine 1.3% or Bupivacaine-Epinephrine 0.25%, 1:200,000. At the end of surgery, study drug will be administered as per the standard FDA guidelines. Study drug will be administered by the investigator surgeon or members of surgical team under supervision of the investigator surgeon. Dose will be calculated by the surgeon based on the screening weight of each randomized participant as is done as the standard of care. Treatment compliance will be measured in terms of the subject receiving an injection of either Liposomal Bupivacaine 1.3% or Bupivacaine-Epinephrine 0.25%, 1:200,000 from the study personnel. No other forms of compliance will be measured. Reasons for any deviation will be recorded. Outcomes will be measured during post-operative hospital stay and until 1 year after surgery for extended follow up which is the standard protocol with cardiothoracic surgery.

Study coordinators will be responsible for data collection and will ensure that forms are completed and signed. Protected Health Information (PHI) will be recorded for tracking the participants through the course of the study. Subjects may be assigned an identification number for unbiased analysis, and will be linked to PHI separately. Data will be collected on data collection forms and subsequently entered into REDCap. Original signed consent forms, data collection forms and any relevant source documentation will be maintained for the duration of the study in locked file cabinets in the department of Cardiothoracic Surgery, Southern Illinois University, Springfield, IL. Electronic data will be stored on a secure server accessible via password-protected computer. Only authorized study personnel will have access to the study data. After completion of data analysis and final manuscript(s) approval, all non-electronic records will be sent to university records management for extended storage. Records will be stored for such a period after study completion as dictated by the university regulations. Adverse events, serious adverse events, discontinuation of drug administration due to adverse events will monitored for both the study drugs and will be reported to the Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

1. Adult at least 18 years of age
2. Subject needs elective lobectomy for non small cell lung cancer
3. Willing to comply with all aspects of protocol, including providing information about opioid usage for post-surgical pain and signed informed consent

Exclusion Criteria:

1. < 18 years of age, > 80 years of age
2. Inability or unwillingness to consent
3. Emergency surgery
4. Previous ipsilateral thoracic surgery
5. Need for operative pleurectomy or pleurodesis
6. Chronic Narcotic use
7. Any narcotic use in the 1 month period prior to screening
8. Allergies to bupivacaine or other local anesthetics, narcotics, NSAIDs or acetaminophen
9. Moderate to severe hepatic impairment (ALT or AST) value greater than 3 times the upper limit of normal.
10. Severe renal impairment or end stage renal failure disease (creatinine greater than 2.0 mg/dl).
11. History of peptic ulcerative disease
12. Severe chronic obstructive pulmonary disease (COPD) due to LVRS (lung-volume reduction surgery).
13. Pregnancy
14. Need for conversion from a Video-Assisted Thoracic Surgery procedure to an open thoracotomy
15. Subjects who are incarcerated
16. Subject has been treated with an experimental device within 30 days or received an experimental agent within the longer of 30 days or five half-lives. Or subject is current enrolled in another clinical trial.
17. Unable to follow protocol directions due to organic brain or psychiatric disease.
18. History of alcoholism or any other substance abuse, which, in the opinion of the investigator, would affect compliance with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Traves Crabtree, MD, Principal Investigator — Professor of Surgery; Stephen Hazelrigg, MD, Study Director — Professor of Surgery
Locations (1):
- Memorial Medical Center, Southern Illinois University-School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel | Marcaine
Started | 29 | 28
Completed | 26 | 24
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Marcaine | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.6) | 66.5 (7.7) | 66 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 19 | 19 | 38
  Obesity | 7 | 5 | 12
  Diabetes Mellitus | 4 | 7 | 11
  COPD | 5 | 9 | 14
  Asthma | 4 | 1 | 5
  Arthritis | 4 | 1 | 5
  GERD | 8 | 8 | 16
  Hyperlipidemia | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Equivalents Consumed
Description: Measured as overall intake of any drugs in the opioid class (Morphine Equivalent Dosing)
Time Frame: up to 72 hours post surgery
Measure: Median (Inter-Quartile Range); unit: MEq
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
MEq | 48 [23 to 71] | 42.7 [28.4 to 55.5]

2. Secondary Outcome: VAS Pain Score
Description: Using a 10 point visual analog scale (VAS) score. The score ranges from 0 to 10. '0' represents no pain and '10' represents worst pain.
Time Frame: In-hospital until discharge, approximately 3 days, will be collected each time before dispensing pain medications
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
score on a scale | 4.8 [4.3 to 6.2] | 5.2 [4.2 to 6.6]

3. Secondary Outcome: Treatment Cost
Description: All direct cost from the date of surgery until discharge
Time Frame: In-hospital Costs until discharge, approximately 3 days
Measure: Median (Inter-Quartile Range); unit: United States Dollars
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
United States Dollars | 22,775 [19,930 to 30,659] | 20,252 [18,225 to 25,521]

4. Secondary Outcome: Pharmacy Cost
Description: Median In-hospital pharmacy cost
Time Frame: In-hospital until discharge, approximately 3 days
Measure: Median (Inter-Quartile Range); unit: United States Dollars
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
United States Dollars | 1052 [970 to 1295] | 596 [497 to 738]

5. Secondary Outcome: Mortality
Description: Any death occurring during primary hospital stay or prior to 30 days post surgery
Time Frame: Up to 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
Participants | 0 | 0

6. Other Pre Specified Outcome: Hospital Stay
Time Frame: Length of hospital stay - from admission to discharge, approximately 3 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
Days | 3.28 [2.16 to 4.27] | 2.45 [2.08 to 3.45]

7. Other Pre Specified Outcome: Pneumothorax
Description: Documented pnuemothorax
Time Frame: In-hospital until discharge, approximately 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
Participants | 5 | 6

8. Other Pre Specified Outcome: Prolonged Air Leak
Description: Number of patients who had air leak more than 5 days post-surgery
Time Frame: > 5 days to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
Participants | 8 | 5

9. Other Pre Specified Outcome: Atrial Fibrillation/Other Arrhythmia
Description: Post-op arrhythmia
Time Frame: In-hospital until discharge, approximately 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 26 | 24
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 30 days post surgery
Description: Follow-up period for all-cause mortality was 30 days. Any air-lead >5 days to 7 days was documented as Prolonged air leak Follow-up period for all other adverse events was in-hospital until discharge, approximately 30 days.
Arm/Group | Exparel | Marcaine
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 12/26 | 9/24
Other Adverse Events (participants affected / at risk) | 2/26 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel (N=26) | Marcaine (N=24)
Prolonged air leak (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Atrial Fibrillation/Other Arrhythmia (Cardiac disorders) | 2 | 3
Infection (Infections and infestations) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel (N=26) | Marcaine (N=24)
Acute Renal Failure (Renal and urinary disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03682224/Prot_SAP_000.pdf